CLINICAL TRIAL: NCT02517515
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of ABT-450/Ritonavir/ABT-267 (ABT-450/r/ABT-267) and ABT-333 in Treatment-Naïve and Treatment-Experienced, Non-Cirrhotic Asian Adults With Subgenotype 1b Chronic Hepatitis C Virus (HCV) Infection
Brief Title: ABT-450/Ritonavir/ABT-267 (ABT-450/r/ABT-267) and ABT-333 in Treatment-Naïve and Treatment-Experienced, Non-Cirrhotic Asian Adults With Subgenotype 1b Chronic Hepatitis C Virus (HCV) Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M13-767
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Results first posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-09

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: HCV Infection; Chronic Hepatitis C Virus; Hepatitis C Virus (HCV) Genotype 1b
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — ombitasvir; dasabuvir; Viekira Pak; paritaprevir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Double-blind 3-DAA (Experimental): Double-blind 3-DAA (ombitasvir/paritaprevir/ritonavir [25 mg/150 mg/100 mg once daily] and dasabuvir [250 mg twice daily]) for 12 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir
- Double-blind Placebo Followed by Open-label 3-DAA (Experimental): Double-blind placebo for 12 weeks, followed by open-label 3-DAA (ombitasvir/paritaprevir/ritonavir [25 mg/150 mg/100 mg once daily] and dasabuvir [250 mg twice daily]) for 12 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir; Drug: Placebo for ombitasvir/paritaprevir/ritonavir and dasabuvir

INTERVENTIONS:
Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir — Tablet; ombitasvir coformulated with paritaprevir and ritonavir, dasabuvir tablet
  Other Names: Viekira Pak; paritaprevir also known as ABT-450; ombitasvir also known as ABT-267; dasabuvir also known as ABT-333
Drug: Placebo for ombitasvir/paritaprevir/ritonavir and dasabuvir — Placebo for ombitasvir/paritaprevir/ritonavir and dasabuvir
  Arms: Double-blind Placebo Followed by Open-label 3-DAA

SUMMARY:
This is a study to evaluate ABT 450/r/ABT-267 and ABT-333 in treatment-naïve and treatment-experienced Asian adults with subgenotype 1b chronic HCV without cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Chinese, South Korean, and Taiwanese descent with full Chinese, South Korean, and Taiwanese parentage
* Chronic hepatitis C virus (HCV) infection prior to study enrollment.
* Screening laboratory result indicating HCV subtype 1b (GT1b) infection.
* Per local standard practice, documented absence of cirrhosis.
* Participant has never received antiviral treatment (including interferon [IFN]-based therapy [alpha, beta or pegylated (peg)IFN] with or without RBV) for HCV infection (treatment-naïve participant) or participant must have documentation that they met the definition of one of the following categories (treatment experienced participant): Non-responder or Relapser
* Participant has plasma HCV RNA level > 10,000 IU/mL at Screening.

Exclusion Criteria:

* HCV genotype performed during screening indicating unable to genotype or infection with any HCV genotype other than GT1b.
* Positive test result at Screening for hepatitis B surface antigen (HBsAg), or hepatitis B virus DNA (HBV-DNA) > Lower Limit of Quantification (LLOQ) if HBsAg negative, or anti-human immunodeficiency virus antibody (HIV Ab) positive.
* Any current or past clinical evidence of cirrhosis.
* Any primary cause of liver disease other than chronic HCV infection.
* Screening laboratory analyses showing abnormal kidney, hepatic, or hematologic function.
* Use of known strong inducers of cytochrome P450 3A (CYP3A) or strong inhibitors of cytochrome P450 3A (CYP2C8) within 2 weeks or within 10 half-lives, whichever is longer, of the respective medication/supplement prior to study drug administration.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

REFERENCES:
- [Derived] Zha J, Ding B, Wang H, Zhao W, Yu C, Alves K, Mobashery N, Luo Y, Menon RM. Pharmacokinetics of Ombitasvir, Paritaprevir, Ritonavir, and Dasabuvir in Healthy Chinese Subjects and HCV GT1b-Infected Chinese, South Korean and Taiwanese Patients. Eur J Drug Metab Pharmacokinet. 2019 Feb;44(1):43-52. doi: 10.1007/s13318-018-0492-8. PMID 29909549
- See also: Related Info. — http://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Double-blind 3-DAA | Double-blind Placebo Followed by Open-label 3-DAA
Started | 325 | 325
Completed | 323 | 323
Not Completed | 2 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrew Consent | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind 3-DAA | Double-blind Placebo Followed by Open-label 3-DAA | Total
Number analyzed (Participants) | 325 | 325 | 650
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (13.84) | 45.6 (14.05) | 46.2 (13.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 177 | 352
  Male | 150 | 148 | 298

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of active study drug. The primary efficacy endpoint was superiority of the percentage of treatment-naïve and treatment-experienced HCV subgenotype 1b (GT1b)-infected participants treated with 3-DAA (ombitasvir/paritaprevir/ritonavir [25 mg/150 mg/100 once daily] and dasabuvir [250 mg twice daily]) who achieved SVR12 compared with the historical control rate for comparable patients treated with telaprevir (TVR) plus pegylated interferon (pegIFN) and RBV.
Time Frame: 12 weeks after the last actual dose of active study drug
Population: All treatment-naïve and treatment-experienced participants who received at least 1 dose of active study drug; participants with missing data after backward imputation were counted as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Double-blind 3-DAA (Treatment-Naïve): Participants who were treatment-naïve and received double-blind 3-DAA (ombitasvir/paritaprevir/ritonavir [25 mg/150 mg/100 mg once daily] and dasabuvir [250 mg twice daily]) for 12 weeks.
- Double-blind 3-DAA (Treatment-Experienced): Participants who were treatment-experienced and received double-blind 3-DAA (ombitasvir/paritaprevir/ritonavir [25 mg/150 mg/100 mg once daily] and dasabuvir [250 mg twice daily]) for 12 weeks.
Arm/Group | Double-blind 3-DAA (Treatment-Naïve) | Double-blind 3-DAA (Treatment-Experienced)
Number analyzed (Participants) | 184 | 141
percentage of participants | 99.5 [97.0 to 99.9] | 100 [97.4 to 100.0]
Statistical Analysis 1: Comparison: Double-blind 3-DAA (Treatment-Naïve); Based on a 2-sided significance level of 0.05 and an underlying rate of 96% for the Double-blind 3-DAA treatment-naïve group, the sample size 180 treatment-naïve participants provided >90% power to demonstrate superiority of the regimen to the historical rate for treatment-naïve patients treated with TVR + pegIFN + RBV (80%) (based on one-sample chi-square test of a single binomial proportion for superiority); Test type: Superiority — The superiority of the rate of sustained virologic response at 12 weeks after treatment (SVR12) for the treatment-naïve participants in the Double-blind 3-DAA group as compared with the historical rate for treatment-naïve patients treated with TVR + pegIFN + RBV was analyzed; the lower confidence bound of the 2-sided 95% confidence interval (95% CI) for the percentage of participants with SVR12 must exceed 84% to achieve superiority; percentage of participants = 99.5, 95% CI 2-sided [97.0 to 99.9]
Statistical Analysis 2: Comparison: Double-blind 3-DAA (Treatment-Experienced); Based on a 2-sided significance level of 0.05 and an underlying rate of 96% for the Double-blind 3-DAA treatment-experienced group, the sample size 180 treatment-experienced participants provided >90% power to demonstrate superiority of the regimen to the historical rate for treatment-experienced patients treated with TVR + pegIFN + RBV (80%) (based on one-sample chi-square test of a single binomial proportion for superiority); Test type: Superiority — The superiority of the rate of sustained virologic response at 12 weeks after treatment for the treatment-experienced participants in the Double-blind 3-DAA group as compared with the historical rate for treatment-experienced patients treated with TVR + pegIFN + RBV was analyzed; the lower confidence bound of the 2-sided 95% CI for the percentage of participants with sustained virologic response at 12 weeks after treatment must exceed 75% to achieve superiority; percentage of participants = 100, 95% CI 2-sided [97.4 to 100.0]

2. Primary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks Post-treatment (SVR24)
Description: SVR24 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of active study drug. The primary efficacy endpoint was superiority of the percentage of treatment-naïve and treatment-experienced HCV subgenotype 1b (GT1b)-infected participants treated with 3-DAA (ombitasvir/paritaprevir/ritonavir [25 mg/150 mg/100 once daily] and dasabuvir [250 mg twice daily]) who achieved SVR24 compared with the historical control rate for comparable patients treated with telaprevir (TVR) plus pegylated interferon (pegIFN) and RBV.
Time Frame: 24 weeks after the last actual dose of active study drug
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-blind 3-DAA (Treatment-Naïve) | Double-blind 3-DAA (Treatment-Experienced)
Number analyzed (Participants) | 184 | 141
percentage of participants | 99.5 [97.0 to 99.9] | 100 [97.4 to 100.0]
Statistical Analysis 1: Comparison: Double-blind 3-DAA (Treatment-Naïve); [analysis description as in outcome 1, analysis 2]; Test type: Superiority — The superiority of the rate of sustained virologic response at 24 weeks after treatment (SVR24) for the treatment-naïve participants in the Double-blind 3-DAA group as compared with the historical rate for treatment-naïve patients treated with TVR + pegIFN + RBV was analyzed; the lower confidence bound of the 2-sided 95% confidence interval (95% CI) for the percentage of participants with SVR24 must exceed 84% to achieve superiority; percentage of participants = 99.5, 95% CI 2-sided [97.0 to 99.9]
Statistical Analysis 2: Comparison: Double-blind 3-DAA (Treatment-Experienced); [analysis description as in outcome 1, analysis 2]; Test type: Superiority — The superiority of the rate of sustained virologic response at 24 weeks after treatment (SVR24) for the treatment-experienced participants in the double-blind 3-DAA group as compared with the historical rate for treatment-experienced patients treated with TVR + pegIFN + RBV was analyzed; the lower confidence bound of the 2-sided 95% CI for the percentage of participants with SVR24 must exceed 75% to achieve superiority; percentage of participants = 100, 95% CI 2-sided [97.4 to 100.0]

3. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed HCV RNA ≥ LLOQ after HCV RNA < LLOQ during active treatment; confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline in HCV RNA during active treatment; or all on-treatment values of HCV RNA ≥ LLOQ with at least 6 weeks of active treatment.
Time Frame: up to 12 weeks
Population: All participants who received at least 1 dose of active study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-blind 3-DAA (Treatment-Naïve) | Double-blind 3-DAA (Treatment-Experienced)
Number analyzed (Participants) | 184 | 141
percentage of participants | 1.1 [0.3 to 3.9] | 0 [0.0 to 2.7]

4. Secondary Outcome: Percentage of Participants With Post-treatment Relapse by Post-treatment Week 12
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of active study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment.
Time Frame: From the end of treatment through 12 weeks after the last dose of active study drug
Population: All participants who received at least 1 dose of active study drug, completed treatment, and had HCV RNA <LLOQ at the final treatment visit, who had HCV RNA data available during the SVR12 period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-blind 3-DAA (Treatment-Naïve) | Double-blind 3-DAA (Treatment-Experienced)
Number analyzed (Participants) | 183 | 141
percentage of participants | 0 [0.0 to 2.1] | 0 [0.0 to 2.7]

5. Secondary Outcome: Percentage of Participants With Post-treatment Relapse by Post-treatment Week 24
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 24 weeks after the last dose of active study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment.
Time Frame: From the end of treatment through 24 weeks after the last dose of active study drug
Population: All participants who received at least 1 dose of active study drug, completed treatment, and had HCV RNA <LLOQ at the final treatment visit, who had HCV RNA data available during the SVR24 period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-blind 3-DAA (Treatment-Naïve) | Double-blind 3-DAA (Treatment-Experienced)
Number analyzed (Participants) | 183 | 141
percentage of participants | 0 [0.0 to 2.1] | 0 [0.0 to 2.7]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) for the double-blind (DB) period were collected from first dose of DB study drug until 30 days after the last dose of DB study drug or until the first dose of open-label (OL) study drug for those entering the OL period (up to 16 weeks). TEAEs and TESAEs for the OL period were collected from the first dose of OL study drug until 30 days after the last dose of OL study drug (up to 16 weeks).
Groups:
- Double-blind Placebo: Double-blind placebo for 12 weeks.
- Open-label 3-DAA: Open-label 3-DAA (ombitasvir/paritaprevir/ritonavir [25 mg/150 mg/100 mg once daily] and dasabuvir [250 mg twice daily]) for 12 weeks.
Arm/Group | Double-blind 3-DAA | Double-blind Placebo | Open-label 3-DAA
Serious Adverse Events (participants affected / at risk) | 7/325 | 2/325 | 5/324
Other Adverse Events (participants affected / at risk) | 72/325 | 61/325 | 55/324
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind 3-DAA (N=325) | Double-blind Placebo (N=325) | Open-label 3-DAA (N=324)
ANAL FISSURE (Gastrointestinal disorders) | 0 | 1 | 0
CROHN'S DISEASE (Gastrointestinal disorders) | 1 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 0
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 | 0 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 0
CHEST DISCOMFORT (General disorders) | 1 | 0 | 0
LUNG INFECTION (Infections and infestations) | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 1 | 0 | 0
ABORTION INDUCED (Surgical and medical procedures) | 1 | 0 | 0
VARICOSE VEIN (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind 3-DAA (N=325) | Double-blind Placebo (N=325) | Open-label 3-DAA (N=324)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 7 | 18 | 7
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 33 | 29 | 31
DIZZINESS (Nervous system disorders) | 17 | 10 | 9
HEADACHE (Nervous system disorders) | 20 | 13 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.